CLINICAL TRIAL: NCT04849416
Title: A Phase 2 Study of Oral LOXO-305 in Patients With Previously Treated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) or Non-Hodgkin Lymphoma (NHL)
Brief Title: A Study of LOXO-305 in Chinese Participants With Blood Cancer (Including Lymphoma and Chronic Leukemia)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17746; J2N-MC-JZNJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-04-16; First posted 2021-04-19 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-08

CONDITIONS: Leukemia, Lymphoid; Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphoid; Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- LOXO-305 (Experimental): Participants received 200 mg of LOXO-305 administered orally once daily (QD) on Days 1 through 28 of a 28-day cycle. The treatment was continued until progressive disease, a discontinuation criterion, or unacceptable toxicity.
  Interventions: Drug: LOXO-305

INTERVENTIONS:
Drug: LOXO-305 — Administered orally.
  Other Names: LY3527727; Pirtobrutinib

SUMMARY:
A study of the safety, side effects, and effectiveness of LOXO-305 in Chinese adults with lymphoma or chronic leukemia who have already had standard of care treatment. Participation could last up to four years.

ELIGIBILITY:
Inclusion Criteria

* Participants with histologically confirmed B-cell malignancy including:

  * Mantle cell lymphoma (MCL) treated with a prior Bruton's tyrosine kinase (BTK) inhibitor containing regimen;
  * CLL/SLL treated with a prior BTK inhibitor containing regimen;
  * Other types of B-cell NHL
* All participants must have disease requiring treatment, for CLL/SLL participants, at least 1 indication for treatment consistent with IWCLL 2018 criteria is required
* Eastern Cooperative Oncology Group 0-2
* Adequate hematologic status, coagulation, hepatic and renal function

Exclusion Criteria

* Lack of adequate wash-out period for investigational agent or anticancer therapy, major surgery, and radiotherapy prior to the first dose of study treatment
* Participants requiring therapeutic anticoagulation with warfarin
* Known central nervous system (CNS) involvement by systemic lymphoma. Primary CNS lymphoma is excluded
* Significant cardiovascular disease
* Prolongation of the QT interval
* Test positive for human immunodeficiency virus (HIV)
* Current treatment with certain strong cytochrome P450 3A4 (CYP450 3A4) inhibitors or inducers and/or strong p-glycoprotein (P-gp) inhibitors
* Pregnancy or lactation
* Active second malignancy
* Prior treatment with LOXO-305
* Known hypersensitivity to any component or excipient of LOXO-305

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2025-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- China (22):
  - Wannan Medical College Yijishan Hospital, Wuhu, Anhui
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Institute of hematology&blood disease hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Medical University Cancer Hospital - Urumqi, Ürümqi, Xinjiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Shanghai East Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting
Access Criteria: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting
URL: http://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Mantle Cell Lymphoma (MCL) Cohort: Participants with MCL received 200 milligrams (mg) of LOXO-305 administered orally once daily (QD) on Days 1 through 28 of a 28-day cycle. The treatment was continued until progressive disease, a discontinuation criterion, or unacceptable toxicity.
- Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL) Cohort: Participants with CLL or SLL received 200 mg of LOXO-305 administered orally QD on Days 1 through 28 of a 28-day cycle. The treatment was continued until progressive disease, a discontinuation criterion, or unacceptable toxicity.
- Other Cohort: Participants with other B cell non-Hodgkin lymphoma (NHL) received 200 mg of LOXO-305 administered orally QD on Days 1 through 28 of a 28-day cycle. The treatment was continued until progressive disease, a discontinuation criterion, or unacceptable toxicity.
Period: Overall Study
Arm/Group | Mantle Cell Lymphoma (MCL) Cohort | Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL) Cohort | Other Cohort
Started | 39 | 17 | 31
Received At Least One Dose of Study Drug | 39 | 17 | 31
Completed (Completers included participants who died from any cause and who did not attend the Follow-up.) | 18 | 3 | 17
Not Completed | 21 | 14 | 14
Not completed — Ongoing Treatment | 12 | 5 | 3
Not completed — On Post-Treatment Follow-up | 8 | 9 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- MCL Cohort: Participants with MCL who received 200 mg of LOXO-305 administered orally QD. on Days 1 through 28 of a 28-day cycle. The treatment was continued until progressive disease, a discontinuation criterion, or unacceptable toxicity.
- CLL/SLL Cohort: Participants with CLL or SLL who received 200 mg of LOXO-305 administered orally QD on Days 1 through 28 of a 28-day cycle. The treatment was continued until progressive disease, a discontinuation criterion, or unacceptable toxicity.
- Other Cohort: Participants with other B cell NHL who received 200 mg of LOXO-305 administered orally QD on Days 1 through 28 of a 28-day cycle. The treatment was continued until progressive disease, a discontinuation criterion, or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | MCL Cohort | CLL/SLL Cohort | Other Cohort | Total
Number analyzed (Participants) | 39 | 17 | 31 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (7.4) | 60.8 (9.2) | 59.9 (9.9) | 62.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 13 | 31
  Male | 27 | 11 | 18 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 39 | 17 | 31 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 39 | 17 | 31 | 87
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 39 | 17 | 31 | 87

OUTCOME MEASURES:

1. Primary Outcome: Primary Analysis Set (PAS): Overall Response Rate (ORR) Assessed by Independent Review Committee
Description: ORR was assessed by an Independent Review Committee (IRC). It was estimated based on the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR). Two-sided 95% CI was calculated using the exact binomial distribution. PAS consisted of participants with Central histologically confirmed non-blastoid MCL, with no CNS metastases and treated with prior chemoimmunotherapy and BTK inhibitor-containing regimen, measurable disease at baseline as assessed using Lugano criteria, and have received at least 1 dose of study drug.
Time Frame: Date of First Dose to Date of Disease Progression or Subsequent Anti-cancer Therapy (up to 100 Weeks)
Population: All participants with Central histologically confirmed non-blastoid MCL, with no CNS metastases and treated with prior chemoimmunotherapy and BTK inhibitor-containing regimen, measurable disease at baseline as assessed using Lugano criteria, and have received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PAS - MCL Group: Participants received 200 mg of LOXO-305 administered orally QD.
Arm/Group | PAS - MCL Group
Number analyzed (Participants) | 28
Percentage of participants | 71.4 [51.3 to 86.8]

2. Secondary Outcome: PAS ORR: ORR Assessed by Investigator
Description: ORR was assessed by the Investigator. It was estimated based on the percentage of participants with BOR of CR or PR. Two-sided 95% CI was calculated using the exact binomial distribution.
Time Frame: Date of First Dose to Date of Disease Progression or Subsequent Anti-cancer Therapy (up to 100 Weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PAS - MCL Group
Number analyzed (Participants) | 28
Percentage of participants | 64.3 [44.1 to 81.4]

3. Secondary Outcome: PAS Best Overall Response (BOR): Percentage of Participants With CR, PR, Stable Disease (SD), Progressive Disease (PD) or Not Evaluable (NE)
Description: BOR was assessed by the IRC and Investigator. Best overall assessment categories include (in descending order of extent of response): CR, PR, SD, PD, and NE. Two-sided 95% CI was calculated using the exact binomial distribution.
Time Frame: Date of First Dose to Date of Disease Progression or Subsequent Anti-cancer Therapy (up to 100 Weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PAS - MCL Group
Number analyzed (Participants) | 28
Percentage of participants
  CR by IRC | 14.3 [4.00 to 32.7]
  PR by IRC | 57.1 [37.2 to 75.5]
  SD by IRC | 7.1 [0.9 to 23.5]
  PD by IRC | 14.3 [4.0 to 32.7]
  NE by IRC | 7.1 [0.9 to 23.5]
  CR by Investigator | 14.3 [4.0 to 32.7]
  PR by Investigator | 50.0 [30.7 to 69.4]
  SD by Investigator | 10.7 [2.3 to 28.2]
  PD by Investigator | 17.9 [6.1 to 36.9]
  NE by Investigator | 7.1 [0.9 to 23.5]

4. Secondary Outcome: PAS: Duration of Response (DOR)
Description: DOR was assessed by the Investigator and IRC. DOR is defined as the number of months from the date of the first documented response to the date of PD or death, whichever occurs earlier. Participants who are alive and without documented PD as of data analysis cutoff date will be censored.
Time Frame: Date of CR or PR to Date of Disease Progression or Death Due to Any Cause (Up to 100 Weeks)
Population: All eligible participants who had Central histologically confirmed non-blastoid MCL with no CNS metastases and treated with prior chemoimmunotherapy and BTK inhibitor-containing regimen, had measurable disease at baseline as assessed using Lugano criteria and received at least 1 dose of study drug with response. Number of participants censored for IRC assessment:13. Number of participants censored for Investigator assessment:8.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PAS - MCL Group
Number analyzed (Participants) | 20
Months
  IRC Assessment | NA [4.83 to NA] — Median and upper limit of the 95% Confidence Interval (CI) was not evaluable because there were insufficient number of participants with events.
  Investigator Assessment: number analyzed (Participants) | 18
  Investigator Assessment | 11.50 [3.68 to NA] — The upper limit of 95% CI was not evaluable because there were insufficient number of participants with events

5. Secondary Outcome: PAS: Progression Free Survival (PFS)
Description: PFS was assessed by the IRC and Investigator. PFS is defined as the number of months from the date of the first dose of study drug to the earlier of documented PD or death due to any cause. Participants who are alive and without documented PD as of data analysis cutoff date were censored.
Time Frame: Date of First Dose to Progressive Disease or Death from Any Cause (Up to 100 weeks)
Population: All eligible participants who had Central histologically confirmed non-blastoid MCL with no CNS metastases and treated with prior chemoimmunotherapy and BTK inhibitor-containing regimen, had measurable disease at baseline as assessed using Lugano criteria and received at least 1 dose of study drug. Number of participants censored for IRC assessment: 15. Number of participants censored for Investigator assessment: 10.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- PAS - MCL Group: Participants received 200 mg of LOXO-305 administered orally QD. Participants included those who had Central histologically confirmed non-blastoid MCL with no CNS metastases and treated with prior chemoimmunotherapy and BTK inhibitor-containing regimen, had measurable disease at baseline as assessed using Lugano criteria and received at least 1 dose of study drug.
Arm/Group | PAS - MCL Group
Number analyzed (Participants) | 28
Months
  IRC Assessment | 9.43 [5.32 to NA] — Upper limit CI was not evaluable because there were insufficient number of participants with events.
  Investigator Assessment | 6.80 [3.61 to 13.34]

6. Secondary Outcome: PAS: Overall Survival (OS)
Description: OS is defined as the number of months elapsed between the date of the first dose of study drug and the date of death from any cause. Participants who are alive or lost to follow-up as of the data cutoff date will be censored.
Time Frame: Date of First Dose to Date of Death from Any Cause (Up to 100 weeks)
Population: All eligible participants who had Central histologically confirmed non-blastoid MCL with no CNS metastases and treated with prior chemoimmunotherapy and BTK inhibitor-containing regimen, had measurable disease at baseline as assessed using Lugano criteria and received at least 1 dose of study drug. Number of participants censored: 16.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PAS - MCL Group
Number analyzed (Participants) | 28
Months | 15.47 [8.67 to NA] — Upper limit CI was not evaluable because there were insufficient number of participants with events.

7. Secondary Outcome: Pharmacokinetics (PK): Area Under the Plasma Concentration Versus Time Curve From Time Zero to Last Quantifiable Concentration(AUC[0-tlast] of LOXO-305
Description: PK: AUC[0-tlast] of LOXO-305
Time Frame: Cycle 1 Day 1: Predose, 1, 2, 4, 8, 12, 24 hours(h) postdose; Cycle 1 Day 8: Predose, 1, 2, 4, 8, 24 h postdose; Cycle 2 Day 1: Predose, 1, 2, 4, 8, 24 h postdose; Cycle 4 Day 1: Predose, 1, 2, 4, 8 h postdose.
Population: All participants who received at least one dose of study drug and had evaluable intensive PK data per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour per milliliter (ng*h/mL)
Groups:
- 200 mg LOXO-305 QD: Participants received 200 mg of LOXO-305 administered orally QD on Days 1 through 28 of a 28-day cycle.
Arm/Group | 200 mg LOXO-305 QD
Number analyzed (Participants) | 13
nanogram hour per milliliter (ng*h/mL)
  Cycle 1 Day 1 | 62700 (15.0)
  Cycle 1 Day 8: number analyzed (Participants) | 12
  Cycle 1 Day 8 | 123000 (38.1)
  Cycle 2 Day 1: number analyzed (Participants) | 11
  Cycle 2 Day 1 | 137000 (28.7)
  Cycle 4 Day 1: number analyzed (Participants) | 12
  Cycle 4 Day 1 | 46600 (20.0)

8. Secondary Outcome: PK: Maximum Concentration (Cmax) of LOXO-305
Description: PK: Cmax of LOXO-305
Time Frame: as for outcome 7
Population: All participants who received at least one dose of study drug and had evaluable intensive PK data per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 200 mg LOXO-305 QD
Number analyzed (Participants) | 13
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1 | 4800 (14.7)
  Cycle 1 Day 8: number analyzed (Participants) | 12
  Cycle 1 Day 8 | 8380 (35.3)
  Cycle 2 Day 1: number analyzed (Participants) | 11
  Cycle 2 Day 1 | 9080 (22.3)
  Cycle 4 Day 1: number analyzed (Participants) | 12
  Cycle 4 Day 1 | 7890 (22.5)

9. Secondary Outcome: PAS: Change From Baseline in Disease-Related Symptoms and Health-Related Quality of Life (HRQoL) Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30 v3.0 was a self-administered questionnaire with multidimensional scales that measures global health status, 5 functional domains (physical, role, cognitive, emotional, and social) and symptom scales of fatigue, pain, nausea and vomiting, dyspnea, loss of appetite, insomnia, constipation, diarrhea, and financial difficulties. A linear transformation is applied to standardize the raw scores to range between 0 and 100 per developer guidelines. For functional domains and global health status, scores range from 0 to 100 with higher scores representing a better level of functioning. For symptoms scales, scores range from 0 to 100 with higher scores representing a greater degree of symptoms.
Time Frame: Baseline, 7 Days After Treatment Discontinuation (Up To 100 Weeks)
Population: All participants who had Central histologically confirmed non-blastoid MCL with no CNS metastases and treated with prior chemoimmunotherapy and BTK inhibitor-containing regimen, had measurable disease at baseline as assessed using Lugano criteria and received at least 1 dose of study drug and EORTC QLQ-C30 data.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | PAS - MCL Group
Number analyzed (Participants) | 27
score on a scale
  Global health status | 2.5 (4.78)
  Functional scale: Physical functioning | 0.8 (2.96)
  Functional scale: Role functioning | -2.9 (3.57)
  Functional scale: Emotional functioning | -2.0 (1.68)
  Functional scale: Cognitive functioning | -1.0 (1.73)
  Functional scale: Social functioning | -7.8 (3.81)
  Symptom scale: Fatigue | -1.3 (3.80)
  Symptom scale: Nausea and vomiting | 0.0 (1.43)
  Symptom scale: Pain | -3.9 (2.27)
  Symptom scale: Dyspnea | -2.0 (1.96)
  Symptom scale: Insomnia | 2.0 (3.47)
  Symptom scale: Appetite loss | -2.0 (4.49)
  Symptom scale: Constipation | -3.9 (2.68)
  Symptom scale: Diarrhea | 0.0 (0.00)
  Symptom scale: Financial difficulties | 3.9 (4.85)

ADVERSE EVENTS:
Time Frame: Baseline Up To 100 Weeks
Description: All participants who received at least one dose of study drug. Per protocol, Adverse Event analysis was planned as per treatment regimen received.
Groups:
- 200 mg LOXO-305 QD: Participants received 200 mg of LOXO-305 administered orally QD on Days 1 through 28 of a 28-day cycle. The treatment was continued until progressive disease, a discontinuation criterion, or unacceptable toxicity.
Arm/Group | 200 mg LOXO-305 QD
All-Cause Mortality (participants affected / at risk) | 37/87
Serious Adverse Events (participants affected / at risk) | 33/87
Other Adverse Events (participants affected / at risk) | 81/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg LOXO-305 QD (N=87)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2)
Covid-19 (Infections and infestations) | 3 (3)
Covid-19 pneumonia (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Pneumonia viral (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Haemorrhage (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg LOXO-305 QD (N=87)
Anaemia (Blood and lymphatic system disorders) | 27 (41)
Leukocytosis (Blood and lymphatic system disorders) | 8 (10)
Leukopenia (Blood and lymphatic system disorders) | 6 (21)
Neutropenia (Blood and lymphatic system disorders) | 10 (32)
Sinus tachycardia (Cardiac disorders) | 6 (6)
Ventricular extrasystoles (Cardiac disorders) | 8 (12)
Abdominal distension (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 11 (14)
Vomiting (Gastrointestinal disorders) | 5 (5)
Asthenia (General disorders) | 5 (6)
Oedema peripheral (General disorders) | 5 (5)
Pyrexia (General disorders) | 13 (16)
Covid-19 (Infections and infestations) | 14 (14)
Pneumonia (Infections and infestations) | 9 (14)
Upper respiratory tract infection (Infections and infestations) | 8 (9)
Urinary tract infection (Infections and infestations) | 7 (8)
Alanine aminotransferase increased (Investigations) | 9 (12)
Aspartate aminotransferase increased (Investigations) | 14 (20)
Bilirubin conjugated increased (Investigations) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 8 (9)
Blood bilirubin increased (Investigations) | 20 (39)
Blood creatinine increased (Investigations) | 11 (22)
Blood lactate dehydrogenase increased (Investigations) | 13 (20)
Gamma-glutamyltransferase increased (Investigations) | 6 (9)
Lymphocyte count decreased (Investigations) | 7 (7)
Neutrophil count decreased (Investigations) | 26 (43)
Platelet count decreased (Investigations) | 13 (17)
Weight increased (Investigations) | 10 (11)
White blood cell count decreased (Investigations) | 19 (39)
Decreased appetite (Metabolism and nutrition disorders) | 5 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (24)
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 (15)
Hyperuricaemia (Metabolism and nutrition disorders) | 17 (27)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (11)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (10)
Hypochloraemia (Metabolism and nutrition disorders) | 7 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 20 (30)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Haematuria (Renal and urinary disorders) | 6 (11)
Proteinuria (Renal and urinary disorders) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 10 (11)
Hypertension (Vascular disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT04849416/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT04849416/SAP_001.pdf